CLINICAL TRIAL: NCT05195424
Title: Estimation of Central Venous Pressure by Echocardiography in Intubated Children in Pediatric Intensive Care: a Prospective Multicenter Study
Brief Title: Estimation of Central Venous Pressure by Echocardiography in Intubated Children in Pediatric Intensive Care
Acronym: PVCECHO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP21
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2021-09

CONDITIONS: Echocardiography in Intubated Children in Pediatric Intensive Care; Intubation Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Estimation of central venous pressure by echocardiography in intubated children in pediatric intensive care — Estimation of central venous pressure by echocardiography in intubated children in pediatric intensive care

SUMMARY:
Central venous pressure (CVP) is a parameter used very regularly in pediatric resuscitation units. According to international recommendations, it should be measured during resuscitation of acute circulatory failure, severe head trauma, renal transplantation in low weight children, or to indirectly assess systolic pulmonary artery pressure by the tricuspid leak gradient. The baseline measurement should be performed using a central venous catheter placed at the right atrial outlet. However, in clinical practice, trans-thoracic echocardiography (TTE) is the most widely used hemodynamic examination in PRU because of its simplicity of use and the excellent echogenicity of patients. While this technique allows assessment of CVP in spontaneously ventilated adults, it is not recommended in positively ventilated adults. Similarly, no pediatric study has formally demonstrated that TTE parameters allow reliable estimation of CVP in mechanically ventilated children, who represent a significant proportion of patients hospitalized in PRUs. The investigators therefore propose to validate TTE assessment of CVP in children on MV in PRU.

The investigators wish to carry out a prospective, non-interventional study over 12 months in 6 pediatric intensive care units in France. The main objective will be to study the correlation between the measurement of the collapsibility index, the distensibility index of the inferior vena cava and the ratio of the maximum diameter of the IVC to the diameter of the abdominal aorta with the measurement of the CVP.

When a patient meets the inclusion criteria, oral information and a paper record will be given to the parental authority holders by the investigator or a physician representing the investigator. After a reflection period of at least 3 hours, the non-objection will be sought and noted in the file. The patient will then be managed according to standard ICU care. The CVP measurements and ultrasound parameters, collected as part of the study, must be carried out in succession, without modifying the ventilator settings or the current therapies.

The first step will be to measure the CVP on 3 occasions, at 30 second intervals, checking for the absence of spontaneous respiration or extra systole that has modified the appearance of the curve. The 2nd step will be to perform the cardiac ultrasound with measurements taken 3 times, at 30 second intervals, repositioning the ETT probe each time.

The investigators hypothesize that the cardiac ultrasound allows to estimate the central venous pressure in pediatric patients, intubated and ventilated in positive pressure thanks to the measurement of these parameters. If confirmed, this data would allow validation of CVP estimation via a simple and noninvasive examination in children in VM. Furthermore, according to the recommendations, the examination of CVP via the catheter requires strict criteria on the position of the catheter (in the superior vena cava territory and at the right atrial junction). Estimation of CVP via ultrasound would therefore make it possible to obtain this data in patients whose catheter does not respect the required position, particularly patients with a catheter in the lower territory.

DETAILED DESCRIPTION:
Central venous pressure (CVP) is a parameter used very regularly in pediatric resuscitation units. According to international recommendations, it should be measured during resuscitation of acute circulatory failure, severe head trauma, renal transplantation in low weight children, or to indirectly assess systolic pulmonary artery pressure by the tricuspid leak gradient. The baseline measurement should be performed using a central venous catheter placed at the right atrial outlet. However, in clinical practice, trans-thoracic echocardiography (TTE) is the most widely used hemodynamic examination in PRU because of its simplicity of use and the excellent echogenicity of patients. While this technique allows assessment of CVP in spontaneously ventilated adults, it is not recommended in positively ventilated adults. Similarly, no pediatric study has formally demonstrated that TTE parameters allow reliable estimation of CVP in mechanically ventilated children, who represent a significant proportion of patients hospitalized in PRUs. The investigators therefore propose to validate TTE assessment of CVP in children on MV in PRU.

The investigators wish to carry out a prospective, non-interventional study over 12 months in 6 pediatric intensive care units in France. The main objective will be to study the correlation between the measurement of the collapsibility index, the distensibility index of the inferior vena cava and the ratio of the maximum diameter of the IVC to the diameter of the abdominal aorta with the measurement of the CVP.

When a patient meets the inclusion criteria, oral information and a paper record will be given to the parental authority holders by the investigator or a physician representing the investigator. After a reflection period of at least 3 hours, the non-objection will be sought and noted in the file. The patient will then be managed according to standard ICU care. The CVP measurements and ultrasound parameters, collected as part of the study, must be carried out in succession, without modifying the ventilator settings or the current therapies.

The first step will be to measure the CVP on 3 occasions, at 30 second intervals, checking for the absence of spontaneous respiration or extra systole that has modified the appearance of the curve. The 2nd step will be to perform the cardiac ultrasound with measurements taken 3 times, at 30 second intervals, repositioning the ETT probe each time.

The investigators hypothesize that the cardiac ultrasound allows to estimate the central venous pressure in pediatric patients, intubated and ventilated in positive pressure thanks to the measurement of these parameters. If confirmed, this data would allow validation of CVP estimation via a simple and noninvasive examination in children in VM. Furthermore, according to the recommendations, the examination of CVP via the catheter requires strict criteria on the position of the catheter (in the superior vena cava territory and at the right atrial junction). Estimation of CVP via ultrasound would therefore make it possible to obtain this data in patients whose catheter does not respect the required position, particularly patients with a catheter in the lower territory.

ELIGIBILITY:
Inclusion Criteria:

* Newborns and children from 2 days post term to 12 years Mechanical ventilation
* Carriers of a central venous catheter in the superior vena cava and ending in the right atrium"

Exclusion Criteria:

-

Ages: 2 Days to 12 Years | Sex: All
Age Groups: Child
Study Population: Intubated pediatric patients in an PICU
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-11-03 (Estimated); Study Completion 2022-11-03 (Estimated)

PRIMARY OUTCOMES:
The correlation between the measurement of the Collapsibility Index, the Distensibility Index of the inferior vena cava and the ratio of the maximum diameter of the IVC to the diameter of the Abdominal Aorta with the measurement of the CVP. | 1 day
  Correlation coefficient value between CI, DI, and IVC dmax /AO measurements and reference method CVP measurement

CONTACTS AND LOCATIONS:
Overall Officials: Perrine SEE, MD, Principal Investigator — Assistace Publique Hopitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] See P, Hayotte A, Le Roux E, Guilbert AS, Collignon C, Denante S, Klifa R, Rambaud J, Brissaud O, Dauger S. Estimation of Central Venous Pressure Using Cardiac Ultrasound of Inferior Vena Cava in Ventilated Children: A Prospective Multicenter Observational Study, 2021-2023. Pediatr Crit Care Med. 2025 Dec 1;26(12):e1421-e1426. doi: 10.1097/PCC.0000000000003834. Epub 2025 Sep 29. PMID 41020643